CLINICAL TRIAL: NCT06460025
Title: Slough in Acute or Chronic Wounds for the Diagnosis of Microbiology Cultivation
Brief Title: Compare Wound Sampling Methods Efficacy in Microbiology Culture
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Head of Wound Healing Center, Peking University Third Hospital
Other Study IDs: Long2024-slough vs. swap
Record Dates: First submitted 2024-05-26; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Microbial Colonization; Infected Wound; Slough
Keywords: Microbial Colonization; Infected Wound; Slough; Biofilm; Sampling
MeSH Terms: conditions — Communicable Diseases; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- slough: slough as the wound specimen for microbiology cultivation
- swap: swap as the wound specimen for microbiology cultivation

SUMMARY:
Slough was a visible indicator of biofilm, which was the most available specimen from acute and chronic wounds. However, studies believed that slough were poorly accurate, and that the Levine swab was more recommended for sampling bacterial culture. This study aimed to compare slough with swab sample and analyze the consistency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute and chronic wounds who were first seen at the Wound Care Centre of Peking University Third Hospital from October 2022 to October 2023;
2. Patients who have followed the wound sample collection SOP to simultaneously take wound swabs and putrefactive samples and send them for bacterial culture;;
3. Patients aged 18 years or older;

Exclusion Criteria:

1. Patients who had been taken only one of the wound samples, either swab or slough;
2. The swab collection did not meet the deifinitions for the exudate method or the Levine technique；
3. Bacterial culture profile was incomplete didn't meet the requirement of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a single-center, retrospective, cross-sectional study, including 131 patients with acute or chronic wounds treated in Wound Healing Center of Peking University Third Hospital from October 2022 to October 2023
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
cohen's k coefficient of Gram Stain between Slough and Swap Specimens | Day 0, patients' the first site in wound healing center
  compare the difference of Gram Stain after bacterial culture between Slough and Swap Specimens, by using statistics of cohen's k coefficient，values of κ from The κ coefficients in 0.81 to 1 waeres interpreted as excellentalmost perfect concordance, with 0.61 to 0.80 asrepresented substantial, 0.41 to 0.60 as mean moderate, 0.21 to 0.40 as fair, and 0 to 0.20 as slight.

SECONDARY OUTCOMES:
cohen's k coefficient of Common pathogens between Slough and Swap Specimens | Day 0, patients' the first site in wound healing center
  compare the difference of Common pathogens after bacterial culture between Slough and Swap Specimens, by using statistics of cohen's k coefficient，values of κ from The κ coefficients in 0.81 to 1 waeres interpreted as excellentalmost perfect concordance, with 0.61 to 0.80 asrepresented substantial, 0.41 to 0.60 as mean moderate, 0.21 to 0.40 as fair, and 0 to 0.20 as slight.
agreements in microbiology cultivation between slough and swap | Day 0, patients' the first site in wound healing center
  compare the agreement of pathogens after bacterial culture between Slough and Swap Specimens, by percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Cai M, Li N, Zhang H, Huang E, Zhao J, Jin M, Zhang L. The value of slough in wounds for the diagnosis of microbiology cultivation. Wound Repair Regen. 2025 Jan-Feb;33(1):e70002. doi: 10.1111/wrr.70002. PMID 39924720